CLINICAL TRIAL: NCT05479396
Title: Study of the Predictive Capacity of Peripheral Muscle Function on Quality of Life Impairment at 1 Year in Subjects With Obesity. A Cohort Study.
Brief Title: The Predictive Capacity of Peripheral Muscle Function on Quality of Life Impairment at 1 Year in Subjects With Obesity
Acronym: OBLITAM
Status: Completed | Type: Observational
Sponsor: Hopital Forcilles (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-A00132-41
Record Dates: First submitted 2022-07-15; First posted 2022-07-29 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-02

CONDITIONS: Obesity
Keywords: muscle assessment; ultrasonography; quality of live
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The assessment of health status and physical function is fundamental in patients with obesity, as they play an important role among the various factors influencing quality of life in this population. Several studies have shown an association between high BMI values and a significant deterioration in quality of life, especially in women. Excess body fat in obese patients appears to be responsible for impaired muscle function. This causal link is probably linked to dysfunctions in adipose tissue, leading to a decrease in the expression of proteins responsible for muscle contraction. The recent literature highlights an alteration in quality of life, particularly in obese and elderly subjects, for which changes in muscle function are partly responsible.

Changes in muscle function can be assessed by simple, rapid and non-invasive tools. These changes in the obese patient could be predictive of reduced quality of life. To our knowledge, no study has evaluated the predictive capacity of muscle alteration assessed by ultrasound on the medium-term quality of life of obese patients.

The main objective of this study is to evaluate the predictive capacity of structural alteration of the quadriceps on the decrease in quality of life at 1 year in patients with obesity.

The secondary objectives are to assess the association between :

* Grip strength and quality of life at 1 year;
* Quadriceps muscle strength and quality of life at 1 year;
* Ultrasound measurements of the quadriceps and quality of life at 1 year;
* Ultrasound measurements of the quadriceps and autonomy at 1 year;
* Grip strength and autonomy at 1 year.

This is a prospective, monocenter, observationnal and cohort study.

All outpatients for nutrition assessment will be included.

DETAILED DESCRIPTION:
1. Rationale 1.1 Obesity, a global public health Obesity is a disease of multifactorial origin, linked to nutritional alterations, genetic, psychological, socio-economic factors and more sedentary behaviour. The prevalence of obesity continues to increase in all age groups and in all socio-economic groups.

1.2. Quality of life: patients with obesity with or without metabolic disorders have impaired health, including mental problems and reduced quality of life. In younger obese subjects,the investigators also observe a decrease in quality of life compared to normal weight subjects, where muscle capacity may be a potential factor associated with impaired quality of life.

1.2.1 Peripheral muscle damage: a decrease in the specific strength of the muscle, a decrease in the strength in relation to the cross-sectional area, is observed in subjects suffering from obesity. There is therefore probably a structural alteration of the muscle in the obese patient, which has not yet been described in the literature. The quantity of muscle fibres decreases and is replaced by the infiltration of adipose and fibrous tissue. This replacement of skeletal muscle fibres decreases muscle quality and increases density, thus altering its function. The reduction in muscle mass relative to fat mass, results in a relative loss of muscle strength available to support and move body weight.

1.3 Peripheral muscle ultrasound: Muscle characteristics, in particular muscle size and quality, have been shown to be related to muscle strength and power as well as cardiovascular performance. Ultrasound can also measure muscle echogenicity. The echogenicity of a B-mode (2D) ultrasound image is expressed by a grey scale. On an ultrasound image, the muscle bundles appear as hypoechoic areas, while the aponeuroses are hyperechoic. In the case of atrophied muscles, represented by hyperechoic structures, there is a decrease in the ability of ultrasound to penetrate deep into the tissue.

2 Research hypothesis The investigators hypothesise that impaired peripheral muscle function is a prognostic factor for impaired quality of life at 1 year in subjects with obesity.

3 Objective 3.1 Main objective The main objective of this study is to evaluate the predictive capacity of structural alteration of the quadriceps on the decrease in quality of life at 1 year in patients with obesity.

3.2 Secondary objectives

The secondary objectives are to assess the association between :

* Grip strength and quality of life at 1 year;
* Quadriceps muscle strength and quality of life at 1 year;
* Ultrasound measurements of the quadriceps and quality of life at 1 year;
* Grip strength and independence at 1 year ;
* Quadriceps muscle strength and autonomy at 1 year;
* Ultrasound measurements of the quadriceps and autonomy at 1 year.

  4. Type of study:This is a prospective, monocenter, obversational cohort study. The research will be conducted in accordance with the protocol.

  5. The duration of recruitment will be 10 months.

  6. Standard assessment procedures: Hand Grip Force, Maximum Voluntary Force of the quadriceps.

  7. Assessment procedures added by the research: Muscle ultrasound, Quality of Life Scale, ADL - The Katz Scale

  8. Statistical aspects: Descriptive statistics will be based on means (+/- standard deviation) or medians [interquartile range] depending on the distribution of quantitative variables. Qualitative variables will be described in terms of numbers and percentages. Univariate comparisons will use the usual statistical tests after verification of the distribution of the variables (Chi2 or Fisher's test, t-test, anova or their non-parametric equivalents Wilcoxon and Kruskal-Wallis tests).

The tests will be performed at the 5% significance level. The 95% confidence intervals will be provided for each estimate.

Calculations will be made using IBM SPSS v21 and R software (version 3.6.1, www.R-project.org).

9 Specific analyses 9.1 Estimation of predictive capacity The occurrence of the event (alteration of quality of life at 1 year) will thus be defined for each of the summary scores (MCS and PCS) and for each of the scores of each SF-36 scale. This will allow the calculation of the AUC of the ROC curves as well as the identification of threshold values of the echogenicity of the femoral rectus allowing the prediction of the occurrence of the alteration in the quality of life.

9.2 Measurement of associations

Measures of association will be made between quality of life and quality of life impairment at 1 year and :

* Grip strength ;
* Quadriceps muscle strength;
* Ultrasound measurements of the quadriceps.

The association measures will be carried out between autonomy and loss of autonomy at 1 year and :

* Grip strength ;
* Quadriceps muscle strength;
* Ultrasound measurements of the quadriceps. Loss of autonomy at 1 year will be defined by a decrease of at least 0.5 points (MCID) on the Katz ADL scale (32).

Measures of association between quantitative variables will be made using Pearson's or Spearman's correlation coefficients depending on the distribution of the data. Measures of association between qualitative variables will be performed using the Chi-square or Fisher test depending on the distribution of the data.

The agreement between quantitative variables will be evaluated using the Bland-Altman method and that between qualitative variables using the Kappa coefficient.

10. Expected results in terms of scientific and professional advances This study will make it possible to evaluate the predictive capacity of muscle function on the alteration of quality of life in patients with obesity hospitalised in HDJ Nutrition. It will also characterise peripheral muscle function and its association with quality of life and autonomy at 1 year, which are not yet clear in the scientific literature. If necessary, these results will make it possible to propose non-invasive and inexpensive predictive tools.

11. Expected benefits for the patient The use of non-invasive muscle function tests could allow early identification of obese subjects at risk of deterioration in quality of life, stratify the risk, and propose an adapted therapeutic strategy, such as the implementation of muscle strengthening and therapeutic education programmes.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients assessment Nutrition
* Obese patients (BMI > 30);
* Patient at least 18 years old at the time of inclusion;
* Affiliation with a social security scheme or beneficiary of such a scheme ;
* Oral, free, informed and express consent of the patient.

Exclusion Criteria:

* Patient's refusal to participate in the study ;
* Known pregnancy ;
* Patient whose state of consciousness is not compatible with obtaining consent ;
* Person subject to a legal protection measure ;
* Patient under guardianship or curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients assessment nutrition will be recruited prospectively and consecutively
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Evaluate the predictive capacity of structural alteration of the quadriceps on the decrease in quality of life at 1 year in patients with obesity | Through study completion, an average of 22 months
  The main outcome is the predictive ability of the femoral rectus muscle echogenicity in the gray scale on the 36-Item Short Form Survey (SF-36) score at 1 year

SECONDARY OUTCOMES:
Association between grip strength and quality of life at 1 year | Through study completion, an average of 22 months
  The main outcome is the association between grip strength measured by the hand-grip and the 36-Item Short Form Survey (SF-36) score at 1 year
Association between quadriceps muscle strength and quality of life at 1 year | Through study completion, an average of 22 months
  The main outcome is the association between lower limb strength measured by maximal voluntary quadriceps force dynamometry and the 36-Item Short Form Survey (SF-36) score at 1 year
Association between ultrasound measurements of the quadriceps and quality of life at 1 year | Through study completion, an average of 22 months
  The main outcome is association between ultrasound measurements of the rectus femoris (thickness and mCSA) and the 36-Item Short Form Survey (SF-36) score at 1 year
Association between grip strength and independence at 1 year | Through study completion, an average of 22 months
  The main outcome is the association between grip strength measured by the hand-grip and the Katz Index of Independence in Activities of Daily Living score at 1 year.
  (SCORING: 6 = High (patient independent) 0 = Low (patient very dependent)
Association between quadriceps muscle strength and autonomy at 1 year | Through study completion, an average of 22 months
  The main outcome is the association between lower limb strength measured by maximum voluntary quadriceps force with dynamometry and the Katz Index of Independence in Activities of Daily Living score at 1 year.
  (SCORING: 6 = High (patient independent) 0 = Low (patient very dependent)
Association between ultrasound measurements of the quadriceps and autonomy at 1 year | Through study completion, an average of 22 months
  The main outcome is the association between ultrasound measurements of the rectus femoris (thickness and mCSA) and the Katz Index of Independence in Activities of Daily Living score at 1 year.
  (SCORING: 6 = High (patient independent) 0 = Low (patient very dependent)

CONTACTS AND LOCATIONS:
Overall Officials: Sophie VIDAL-JESSEL, MD, Study Director — Hopital Forcilles; Andreia GOMES LOPES, MSc, Principal Investigator — Hopital Forcilles; Aymeric Le Neindre, Study Chair — Hopital Forcilles
Locations (1):
- Hôpital Forcilles, Férolles-Attilly, France

IPD SHARING:
Plan to Share IPD: Yes
The protocole, the statistical analysis plan and data will be available as supplementary materials with the publication. The other data that support the findings of this study will be available from the corresponding author upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: At publication for 10 years
Access Criteria: The data that support the findings of this study will be available from the corresponding author upon reasonable request.

REFERENCES:
- [Background] Tamura LS, Cazzo E, Chaim EA, Piedade SR. Influence of morbid obesity on physical capacity, knee-related symptoms and overall quality of life: A cross-sectional study. Rev Assoc Med Bras (1992). 2017 Feb;63(2):142-147. doi: 10.1590/1806-9282.63.02.142. PMID 28355375
- [Background] Toselli S, Campa F, Spiga F, Grigoletto A, Simonelli I, Gualdi-Russo E. The association between body composition and quality of life among elderly Italians. Endocrine. 2020 May;68(2):279-286. doi: 10.1007/s12020-019-02174-7. Epub 2019 Dec 31. PMID 31893349
- [Background] Tomlinson DJ, Erskine RM, Winwood K, Morse CI, Onambele GL. The impact of obesity on skeletal muscle architecture in untrained young vs. old women. J Anat. 2014 Dec;225(6):675-84. doi: 10.1111/joa.12248. Epub 2014 Oct 14. PMID 25315680

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-02-22): https://cdn.clinicaltrials.gov/large-docs/96/NCT05479396/Prot_SAP_ICF_000.pdf